CLINICAL TRIAL: NCT04917315
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel, Bridge Study to Evaluate the Efficacy and Safety of JLP-2002 in Patients With Overactive Bladder
Brief Title: To Evaluate the Efficacy and Safety of JLP-2002 on Symptoms of Overactive Bladder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JLP-2002-301
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JLP-2002 (Experimental): Drug: JLP-2002
  Interventions: Drug: JLP-2002 A mg
- Placebo (Placebo Comparator): Drug: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JLP-2002 A mg — administration of JLP-2002 Participants received one vibegron A mg tablet, taken orally each morning, for 12 weeks.
  Arms: JLP-2002
Drug: Placebo — administration of Placebo Participants received one placebo tablet, taken orally each morning, for 12 weeks.
  Arms: Placebo

SUMMARY:
Overactive bladder (OAB) is a clinical condition characterized by urgency (i.e., urinary urinary urinary urgency that is difficult to delay and unbearable) with or without urge incontinence, usually associated with frequency and nocturia. The main drug class used is antimuscarinics, and the clinical utility of antimuscarinic drugs is limited due to its mild efficacy and poor tolerability due to side effects of mechanisms such as dry mouth and constipation. In addition to poor tolerability and mild efficacy, recent literature suggests that long-term use of anticholinergics is associated with cognitive impairment and dementia. Therefore, the purpose of this study was to evaluate the treatment effect of overactive bladder symptoms through the change in the average number of urination per day after administration of JLP-2002, a beta 3-adrenergic receptor (β3-AR) agonist with an effective alternative mechanism, for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Those who are fully informed of this study and then completely understand its contents, voluntarily decide to participate in this study, and give written consent to follow instructions
2. Males or females aged 19 years or older at the time of written consent
3. Those who have already experienced symptoms of overactive bladder (OAB)* for 6 months or more at the time of screening
4. Those who are able to read, understand, and write in a voiding diary and a questionnaire
5. Those who are able to go to the toilet on foot without other's help

Exclusion Criteria:

1. Those who have a history of malignancies within 3 years before screening
2. Those who were previously or are currently diagnosed with urinary malignancies (e.g., bladder cancer)
3. Males who were previously or are currently diagnosed with prostate cancer or whose prostate-specific antigen (PSA) level is ≥ 4ng/mL within 1 year before screening or at screening
4. Those with a history of allergy to β-adrenergic receptor agonists, intolerant or clinically significant adverse events, or abnormal clinical laboratory values
5. Pregnant or lactating women
6. Those whose systolic blood pressure (SBP) is ≥160mmHg; diastolic blood pressure (DBP) is ≥100 mmHg; or pulse is ≥110 bpm at the time of screening and randomization
7. Those who received other investigational products or investigational devices within 30 days before screening
8. Those who are determined by the investigator to be not eligible for this study due to clinically significant abnormal findings of screening tests

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Average Daily Micturitions at Week 12 | Week 12
  Participants were required to keep a voiding diary, recording the occurrence of each micturition. The average daily number of micturitions was calculated as the total number of micturitions that occurred over 3 days during the Base Study, divided by the total number of days of voiding kept in the participant's diary. Baseline was defined as the average daily number of daily micturitions that occurred during the week of placebo run-in prior to Week 0 visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No